CLINICAL TRIAL: NCT02116673
Title: The Influence of Cognitive Rest and Graduated Return to Usual Activities on Minor Traumatic Brain Injury
Brief Title: Influence of Cognitive Rest on Minor Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Catherine Varner, Emergency Physician, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSHED0001
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Minor Head Injury
Keywords: Head injury; Concussion; Cognitive rest; Emergency department
MeSH Terms: conditions — Craniocerebral Trauma; Brain Concussion; Emergencies

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): The control arm receives usual care discharge instructions.
  Interventions: Other: Usual care
- Cognitive rest (Experimental): The intervention is providing discharge instructions instructing cognitive rest and graduated return to usual activities in patients whom have experienced minor traumatic brain injury.
  Interventions: Other: Cognitive rest

INTERVENTIONS:
Other: Cognitive rest — The intervention is providing discharge instructions instructing cognitive rest and graduated return to usual activities in patients whom have experienced minor traumatic brain injury.
  Arms: Cognitive rest
Other: Usual care — These are usual care emergency department discharge instructions provided at emergency department discharge for minor traumatic brain injury.
  Arms: Control

SUMMARY:
Background: Head injury is a common presentation to family medicine clinics and emergency departments (EDs), and the majority will not result in intracranial injury requiring neurosurgical consultation, but will have symptoms of mild traumatic brain injury (MTBI). It is estimated between 15-50% of patients with MTBI develop post-concussive syndrome (PCS). Research in the management of MTBI and prevention of PCS has been scarce to date. Although expert consensus recommends cognitive rest and graduated return to usual activities, these and other interventions are not based on prospective clinical evidence.

Objective: The purpose of this study is to determine if providing graduated return to usual activities discharge instructions to MTBI patients in the ED decreases MTBI symptoms post-injury as compared to providing usual ED MTBI discharge instructions.

Study Design: This will be a pragmatic, single-centered, 2-arm parallel-group, superiority randomized trial.

Patient Population: Male and female patients presenting to the ED ages greater than 17 and less than 65 with the Canadian Emergency Department Information System (CEDIS) presenting complaint of "head injury".

Outcomes: The primary outcome of this study is to determine if patients whom receive graduated return to usual activity discharge instructions have more clinically significant decreases in their Post-Concussion Symptom Score (PCSS) 2 weeks after MTBI versus patients who received usual care MTBI discharge instructions. Secondary outcomes include the intervention group's compliance with the intervention, comparison of PCSS between groups 4 weeks after initial ED visit, comparison of groups' number of return visit(s) to either an ED or physician's office, and the mean number of days of school or work missed for each group.

Hypothesis: Given cognitive rest and graduated return to usual activities are concepts recommended by expert consensus, it is expected patients who follow the graduated return to usual activities and cognitive rest guidelines will have less MTBI symptoms at two weeks after ED discharge.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients presenting to the ED with the Canadian Emergency Department Information System (CEDIS) chief complaint of "head injury".
* Age greater than 17 years and less than 65 years.
* Injury occurring within the last 24 hours.

Exclusion Criteria:

* Acute intracranial injury identified on head CT
* Glasgow Coma Scale (GCS) < 15 at time of discharge
* Non-English speaking

Ages: 17 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Minor traumatic brain injury symptoms | 4 weeks
  Measured by the Post-concussion Symptom Score (PCSS)

SECONDARY OUTCOMES:
Days of work or school missed | 4 weeks
Visits to the emergency department or other health care professionals | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Varner, MD, Principal Investigator — Mount Sinai Hospital Division of Emergency Medicine
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada